CLINICAL TRIAL: NCT02137382
Title: A Double-blind, Randomized, Multicenter, Cross-over Study to Compare the Effect of Creon N and Creon® on Fat Digestion in Subjects ≥ 12 Years of Age With Pancreatic Exocrine Insufficiency Due to Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PANC3004; 2013-002819-10 (EudraCT Number)
Record Dates: First submitted 2014-02-12; First posted 2014-05-13 (Estimated); Results first posted 2015-11-27 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Pancreatic Exocrine Insufficiency Due to Cystic Fibrosis
Keywords: maldigestion of dietary macronutrients (pancreas not producing enough enzymes for digestion of fat, sugars and proteins) in Cystic Fibrosis
MeSH Terms: interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Creon N, then Creon® (Experimental): Subjects first received Creon N for 5 days. After a washout period of 3 to 14 days, they received Creon® for 5 days. The Investigator calculated the total number of capsules per day needed to treat the subject with 8000 to <10000 lipase units per kg body weight and day, Capsules of both Creon N and Creon® contain 25000 lipase units.
  Interventions: Drug: Creon®
- Creon® , then Creon N (Experimental): Subjects first received Creon® for 5 days. After a washout period of 3 to 14 days, they received Creon N for 5 days. The Investigator calculated the total number of capsules per day needed to treat the subject with 8000 to <10000 lipase units per kg body weight and day, Capsules of both Creon N and Creon® contain 25000 lipase units.
  Interventions: Drug: Creon N

INTERVENTIONS:
Drug: Creon® — active comparator
  Arms: Creon N, then Creon®
Drug: Creon N — experimental drug
  Arms: Creon® , then Creon N

SUMMARY:
maldigestion of dietary macronutrients (pancreas not producing enough enzymes for digestion of fat, sugars and proteins) in Cystic Fibrosis

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent given by the subject, or the parents, or a legally acceptable representative. If required by the Institutional Review Board/Ethics Committee (IRB/IEC), assent will be given by the subject
* Age ≥ 12 years
* Subjects who are able to swallow capsules with each meal and snacks
* Diagnosis of Cystic Fibrosis (CF) confirmed by two positive chloride sweat tests or gene analysis
* Diagnosis of pancreatic exocrine insufficiency proven by:

  1. Coefficient of fat absorption (CFA) < 70% without supplementation
  2. or Human fecal elastase < 50 μg/g stool
* Currently receiving treatment with a commercially available pancreatic enzyme product and on a continuous dose of this product for more than 3 months
* Clinically stable condition without evidence of acute respiratory disease within 1 month of enrollment
* Stable body weight defined as no more than a 5% decline within 3 months of enrolment
* Females of child-bearing potential should agree to continue using a medically acceptable method of birth control throughout the study and for 30 days immediately after the last dose of study drug. Medically acceptable methods of birth control include bilateral tubal ligation or the use of either a contraceptive implant, a contraceptive injection (Depo-Provera™), an intrauterine device, or an oral contraceptive taken within the past 3 months where the subject agrees to continue using during the study or to adopt another birth control method, or a double-barrier method which consists of a combination of any two of the following: diaphragm, cervical cap, condom, or spermicide.

Exclusion Criteria:

* Evidence of cardiovascular, respiratory, urogenital, gastrointestinal/hepatic (except underlying disease), hematologic/immunologic, head, ears, eyes, nose, throat, dermatologic/connective tissue, musculoskeletal, metabolic/nutritional (except underlying disease), endocrine (except diabetes mellitus), neurologic/psychiatric, allergy, recent major surgery, or other relevant diseases as revealed by history, physical examination and/or laboratory assessments, which could limit participation in or completion of the study
* History of acute abdomen
* History of fibrosing colonopathy
* History of distal intestinal obstruction syndrome (DIOS) within 6 months prior to enrollment
* Solid organ transplant or surgery affecting the large bowel other than appendectomy
* Small bowel surgery that significantly affected absorptive capacity (e.g. gastrectomy or pancreatectomy)
* Pregnancy or lactation
* Any type of malignancy involving the digestive tract in the last 5 years
* Celiac disease or Crohn's disease
* Known allergy to pancreatin or inactive ingredients (excipients) of pancreatin capsules
* Suspected non-compliance or non-cooperation
* Intake of experimental drugs within 30 days prior to study start
* Mental disability or any other lack of fitness, in the Investigator's opinion, to preclude subject's participation in or ability to complete the study
* Diagnosis of human immunodeficiency virus in medical history.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suntje Sander-Struckmeier, PhD, Study Director — Abbott
Locations (7):
- Hungary (4):
  - Research facility ID ORG-000826, Budapest
  - Research facility ID ORG-000816, Debrecen
  - Research facility ID ORG-000827, Kaposvár
  - Research facility ID ORG-000825, Törökbálint
- Spain (3):
  - Research facility ID ORG-000829, Barcelona
  - Research facility ID ORG-000828, Seville
  - Research facility ID ORG-000815, Valencia

REFERENCES:
- [Derived] Somaraju URR, Solis-Moya A. Pancreatic enzyme replacement therapy for people with cystic fibrosis. Cochrane Database Syst Rev. 2020 Aug 5;8(8):CD008227. doi: 10.1002/14651858.CD008227.pub4. PMID 32761612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 patients consented, between January and March 2014.
Pre-assignment Details: 41 of the 50 patients who consented were randomized; the 9 patients who were not randomized were screening failures.
Groups:
- Sequence: Creon N/Creon®: Subjects first received Creon N for 5 days. After a washout period of 3 to 14 days, they received Creon® for 5 days. The Investigator calculated the total number of capsules per day needed to treat the subject with 8000 to <10000 lipase units per kg body weight and day, Capsules of both Creon N and Creon® contain 25000 lipase units.
- Sequence: Creon®/Creon N: Subjects first received Creon® for 5 days. After a washout period of 3 to 14 days, they received Creon N for 5 days. The Investigator calculated the total number of capsules per day needed to treat the subject with 8000 to <10000 lipase units per kg body weight and day, Capsules of both Creon N and Creon® contain 25000 lipase units.
Period: Cross-over Period 1
Arm/Group | Sequence: Creon N/Creon® | Sequence: Creon®/Creon N
Started | 20 | 21
Completed | 18 | 21
Not Completed | 2 | 0
Period: Wash Out
Arm/Group | Sequence: Creon N/Creon® | Sequence: Creon®/Creon N
Started | 18 | 21
Completed | 18 | 21
Not Completed | 0 | 0
Period: Cross-over Period 2
Arm/Group | Sequence: Creon N/Creon® | Sequence: Creon®/Creon N
Started | 18 | 21
Completed | 18 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence Creon N/Creon® or Creon®/Creon N: Participants who were randomized to receive either Creon N or Creon.
Arm/Group | Sequence Creon N/Creon® or Creon®/Creon N
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 19
Region of Enrollment [Number; unit: Participants]
  Hungary | 15
  Spain | 26

OUTCOME MEASURES:

1. Primary Outcome: Coefficient of Fat Absorption (CFA)
Description: CFA is calculated from fat intake and fat excretion, according to the formula: CFA (%) = 100 [fat intake - fat excretion] / fat intake
Time Frame: 5 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of fat intake
Arm/Group | Creon® | Creon N
Number analyzed (Participants) | 38 | 38
percentage of fat intake | 88.1 (9.23) | 89.5 (6.79)

2. Secondary Outcome: Coefficient of Nitrogen Absorption (CNA).
Description: CNA is calculated from nitrogen intake and nitrogen excretion, according to the formula: CNA (%) = 100 [nitrogen intake - nitrogen excretion] / nitrogen intake)
Time Frame: 5 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of nitrogen intake
Arm/Group | Creon® | Creon N
Number analyzed (Participants) | 38 | 38
percentage of nitrogen intake | 87.7 (5.47) | 87.8 (4.68)

3. Secondary Outcome: Total Fat Excretion
Description: Total amount of fat excreted during the stool collection period in grams.
Time Frame: 5 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Grams
Groups:
- Creon®: Creon® : active comparator
Arm/Group | Creon® | Creon N
Number analyzed (Participants) | 38 | 38
Grams | 48.1 (43.28) | 42.3 (27.05)

4. Secondary Outcome: Stool Frequency
Description: Stool frequency is the average of the daily number of stools recorded during the treatment period
Time Frame: 5 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: number of stools per day
Arm/Group | Creon® | Creon N
Number analyzed (Participants) | 38 | 38
number of stools per day | 1.57 (0.6) | 1.49 (0.6)

5. Secondary Outcome: Percentage of Days With no Flatulence
Description: The percentage of days with no flatulence is calculated from the diary during the treatment period: 100*(number of days with no flatulence/number of days recorded in diary).
Time Frame: 5 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Creon® | Creon N
Number analyzed (Participants) | 38 | 38
percentage of days | 51.6 (46.65) | 57.5 (43.31)

6. Secondary Outcome: Percentage of Days With no Abdominal Pain
Description: The percentage of days with no abdominal pain is calculated from the diary during the treatment period: 100*(number of days with no abdominal pain/ number of days recorded in diary).
Time Frame: 5 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Creon® | Creon N
Number analyzed (Participants) | 38 | 38
percentage of days | 86.8 (22.91) | 89.3 (19.67)

7. Secondary Outcome: Percentage of Days With Formed/Normal Stools
Description: The percentage of days with formed/normal stools is calculated from the diary during the treatment period: 100*(number of days with formed/normal stools/ number of days recorded in diary).
Time Frame: 5 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Creon® | Creon N
Number analyzed (Participants) | 38 | 38
percentage of days | 79.8 (21.21) | 73.6 (29.50)

ADVERSE EVENTS:
Arm/Group | Creon® | Creon N
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41
Other Adverse Events (participants affected / at risk) | 9/39 | 6/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creon® (N=39) | Creon N (N=41)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastro intestinal hyper motility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Steatorrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
viral rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric pH decreased (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No